CLINICAL TRIAL: NCT00697983
Title: Purinergic Signalling in Human Osteoporosis: Evaluation of Variability in Purinergic Receptor Genes and Receptor Function
Brief Title: Cohort Study on Associations Between Purinergic Receptor SNPs and Osteoporosis Risk
Acronym: ATPBone
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Copenhagen University Hospital, Research Center for Aging and Osteoporosis (Unknown); European Commission (Other)
Responsible Party: dr. ir. P.C. Dagnelie, Maastricht University Medical Center
Other Study IDs: MEC 08-3-029; EU FP7, grant no. 202231
Record Dates: First submitted 2008-06-11; First posted 2008-06-16 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; ATP; Purinergic receptors; Bone mineral density; Single nucleotide polymorphism
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fracture cohort: Patients of 50 years and above with a clinical, non-pathological fracture, who attend an osteoporosis outpatient clinic at the Maastricht University Medical Center for standard medical care (including bone densitometry by DXA-scan).

SUMMARY:
Background: Osteoporosis is a high-prevalence disease with a strong genetic component. Nucleotides, including ATP (adenosine 5'-triphosphate) and its purinergic receptors, play a role in bone physiology. Single nucleotide polymorphisms (SNPs) in the P2X7 receptor gene were recently found to be associated with fracture risk in a cohort of postmenopausal women.

Objective: To investigate associations between purinergic receptor SNPs and osteoporosis risk in humans. Genetic data from a fracture cohort in the Netherlands with high prevalence of osteoporosis will be analyzed. Furthermore, effects of aberrant purinergic receptor signalling on bone turnover markers will be assessed ex vivo.

Design: The cohort will include app. 1,000 fracture patients of 50 years and older, who will be recruited at the Maastricht University Medical Center during standard medical follow-up after a clinical fracture. The standard medical follow-up includes assessment of bone mineral density (BMD) by Dual-Energy X-ray Absorptiometry (DXA), if necessary followed by medication for osteoporosis. Prior to medication, blood samples will be collected from fracture patients to be genotyped for purinergic receptor SNPs and analyzed for biochemical markers of bone turnover. Systemic correlates of osteoporosis will be compared between osteoporotic subjects (i.e. low BMD) and non-osteoporotic controls (i.e. normal to high BMD). Subsequently, whole blood assays in patient subgroups (n=20 per subgroup), based on BMD and purinergic receptor SNPs, will be performed to evaluate ex vivo effects of ATP and related nucleotides bone markers.

Study population: Patients of 50 years and older attending an outpatient osteoporosis clinic at the Maastricht University Medical Center for standard medical follow-up after a clinical, non-pathological fracture.

Primary outcome parameters: BMD and purinergic receptor SNPs.

Secondary outcome parameters: Bone markers.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years and older;
* Clinical fracture;
* Attending osteoporosis outpatient clinic for standard medical care.

Exclusion Criteria:

* Disease of bone metabolism (e.g. bone tumours, hyperparathyroidism);
* Unwillingness to donate blood for DNA analyses;
* Failure of bone densitometry (DXA-scan).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fracture patients of 50 years and older attending an osteoporosis outpatient clinic at the Maastricht University Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Purinergic receptor SNPs | cross-sectional
BMD | cross-sectional

SECONDARY OUTCOMES:
Biochemical markers of bone turnover | cross-sectional

CONTACTS AND LOCATIONS:
Overall Officials: Pieter C Dagnelie, PhD, Principal Investigator — Maastricht University, Dept of Epidemiology
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] van Helden S, van Geel AC, Geusens PP, Kessels A, Nieuwenhuijzen Kruseman AC, Brink PR. Bone and fall-related fracture risks in women and men with a recent clinical fracture. J Bone Joint Surg Am. 2008 Feb;90(2):241-8. doi: 10.2106/JBJS.G.00150. PMID 18245581
- [Background] Ohlendorff SD, Tofteng CL, Jensen JE, Petersen S, Civitelli R, Fenger M, Abrahamsen B, Hermann AP, Eiken P, Jorgensen NR. Single nucleotide polymorphisms in the P2X7 gene are associated to fracture risk and to effect of estrogen treatment. Pharmacogenet Genomics. 2007 Jul;17(7):555-67. doi: 10.1097/FPC.0b013e3280951625. PMID 17558311
- [Background] Hoebertz A, Arnett TR, Burnstock G. Regulation of bone resorption and formation by purines and pyrimidines. Trends Pharmacol Sci. 2003 Jun;24(6):290-7. doi: 10.1016/S0165-6147(03)00123-8. PMID 12823955
- [Background] Bours MJ, Swennen EL, Di Virgilio F, Cronstein BN, Dagnelie PC. Adenosine 5'-triphosphate and adenosine as endogenous signaling molecules in immunity and inflammation. Pharmacol Ther. 2006 Nov;112(2):358-404. doi: 10.1016/j.pharmthera.2005.04.013. Epub 2006 Jun 19. PMID 16784779
- [Background] Swennen EL, Bast A, Dagnelie PC. Purinergic receptors involved in the immunomodulatory effects of ATP in human blood. Biochem Biophys Res Commun. 2006 Sep 29;348(3):1194-9. doi: 10.1016/j.bbrc.2006.07.177. Epub 2006 Aug 4. PMID 16904065
- [Background] Bours MJL, Wesselius A en Dagnelie PC. Adenosinetrifosfaat (ATP), purinerge receptoren en botremodellering. Nieuwe perspectieven voor behandeling van osteoporose? Ned Tijdschr Calcium Botstofwisseling 2009; 7(3):71-4.
- See also: European Nucleotides and Bone Consortium — http://www.atpbone.org
- See also: European Commission Research, Seventh Framework Programme — http://ec.europa.eu/research/fp7/index_en.cfm
- See also: University Hospital Maastricht — http://www.azm.nl